CLINICAL TRIAL: NCT06835452
Title: Comparison of Current Subgingival Debridement Methods: Clinical Trial with 6 Months Follow-up
Brief Title: Comparison of Current Subgingival Debridement Methods
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Selcen Ozcan Bulut, Assistant prof, Nigde Omer Halisdemir University
Other Study IDs: 2023/65
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Treatment of Periodontitis; Guided Biofilm Therapy; Subgingival Plaque; Subgingival Debridement
Keywords: guided biofilm therapy; periodontitis; subgingival debridement
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1- classic treatment: Subgingival debridement was performed using the Cavitron and Gracey curette (this is the method that is used routinely).
- Group 2-Guided Biofilm Therapy: Subgingival debridement was performed with the Guided Biofilm Therapy (GBT+Airabrasion) method. This method is the most up-to-date method. The biofilm is shown to the patient with plate dye, and the biofilm is cleaned with air abrasion and perio flow (EMS device cavitron). In the patient's control sessions, the patient's oral hygiene motivation is tried to be increased by dyeing the biofilm.
- Group 3- Classical treatment and with Plaque paint: the dental calculus and biofilm were stained with plaque paint, shown to the patient with the help of a mirror, and then routine subgingival debridement was performed.

SUMMARY:
Our study aimed to compare the effectiveness of current subgingival debridement methods used in the treatment of Stage 1 and Stage 2 periodontitis patients, the aesthetic condition achieved after these treatments, and the pain felt during treatment.

90 female patients who were diagnosed with chronic periodontitis (Stage 1-2) and required supra-subgingival scaling for treatment purposes, and who volunteered to participate in the study, were included in the study. Three treatment groups were determined. 30 people were included in each group. Periodontal examination was performed before and after the treatments in the 1st month, 3rd month and 6th month and the data on the collected periodontal parameters were analyzed.

DETAILED DESCRIPTION:
Periodontal parametreler Gingival index, plaque index, periodontal pocket depth and bleeding index on probing.

It was evaluated with the visual analog scale for pain and aesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patient (without known chronic disease)
* Periodontal diagnostic data (Gingival Index, Plaque Index, Periodontal pocket depths, Attachment loss, Radiological data-Bone loss data) are complete
* Treatments diagnosed with stage 1-2 periodontitis and those who have not had periodontal treatment in the last 6 months

Exclusion Criteria:

* Having a systemic disease
* Pregnant and lactating women
* smoker
* Those who do not want to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 90 female patients with stage 1-2 periodontitis
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Gingival index | baseline, 1st month, 3rd month and 6th month
  4 surfaces of all teeth (distal, buccal, mesial, lingual) are evaluated 0= Normal gingiva
  1. Mild inflammation - slight discoloration, slight edema. There is no bleeding after probing.
  2. Moderate inflammation - redness, edema and shine. Bleeding after probing.
  3. Severe inflammation - marked redness and edema. Ulceration. Tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided